CLINICAL TRIAL: NCT05871541
Title: A Phase 1 Randomized, Double-Blinded, Active-Controlled, 2-Dose Study to Assess the Safety and Immunogenicity of a Herpes Zoster (HZ) Vaccine, JCXH-105, in Healthy Subjects 50 to 69 Years of Age.
Brief Title: A First-in-Human Study to Evaluate JCXH-105, an SrRNA-based Herpes Zoster Vaccine
Acronym: JCXH-105
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immorna Biotherapeutics, Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JCXH-105-001
Record Dates: First submitted 2023-05-03; First posted 2023-05-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-11

CONDITIONS: Herpes Zoster (HZ); Shingles; Infectious Disease
Keywords: srRNA vaccine; Shingles vaccine; Herpes Zoster (HZ) vaccine; Healthy adult participants (aged 50 to 69 years)
MeSH Terms: conditions — Herpes Zoster; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Product (Experimental): Participants randomized to this arm will be given the investigational product (JCXH-105).
  Interventions: Biological: JCXH-105
- Active Control (Active Comparator): Participants randomized to this arm will be given the FDA approved Shingrix.
  Interventions: Biological: Active Control (Shingrix)

INTERVENTIONS:
Biological: JCXH-105 — As IM injection
  Arms: Investigational Product
Biological: Active Control (Shingrix) — As IM injection
  Arms: Active Control

SUMMARY:
The goal of this clinical trial is to assess the safety and immunogenicity of a self-replicating (sr) RNA-based vaccine, JCXH-105, in the prevention of Shingles (Herpes Zoster)

Participant will be randomized to receive either JCXH-105 or Shingrix.

DETAILED DESCRIPTION:
This Phase 1 study plans to enroll a total of 75 participants.

Three cohorts with 3 different dose levels of JCXH-105 will be explored and each cohort will enroll 25 participants (20 randomized to JCXH-105 and 5 randomized to Shingrix) for a total of 75 participants. The dose level of JCXH-105 will depend on the time the participant joins the study. Each participant will receive two single intramuscular (IM) injections of study treatment (JCXH-105 or Shingrix) on day 1 and day 61 (±2 days on day 61)

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male or female; female subjects may be of childbearing potential, of nonchildbearing potential, or postmenopausal.
* Age: 50 to 69 years of age, inclusive, at screening.
* Status: Healthy subjects. Note: Healthy status as defined by the absence of evidence of any clinically significant active or chronic disease, in the opinion of the Investigator, following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG) recording, hematology, blood chemistry, serology, and urinalysis. Healthy subjects may have stable pre-existing disease defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks prior to enrollment.
* Subjects must agree to not be vaccinated with any HZ vaccine while participating in this study.
* All values for hematology and clinical chemistry tests of blood and urine within the normal range OR showing no clinically relevant deviations based on medical history, considering stable pre-existing diseases (see Healthy Subjects above), as judged by the Investigator.

Exclusion Criteria:

* Subjects with a history of HZ or current diagnosis of shingles.
* Previous vaccination against HZ.
* Subjects with any respiratory illness deemed clinically relevant by the Investigator within the past month OR hospitalization >24 hours for any reason within the past month prior to the first vaccine administration (JCXH-105 or Shingrix).
* Subjects with history of myocarditis or pericarditis, or with AEs after mRNA vaccination that are in nature and severity beyond the common expected AEs necessitating medical intervention.
* Subjects who have received an mRNA-based vaccine (e.g., Spikevax, Comirnaty, etc.) 30 days prior to Day 1.
* Subjects who received any non-live vaccine within 14 days prior to the first vaccine administration (JCXH-105 or Shingrix).
* Subjects who received within 28 days prior to first vaccine administration (JCXH-105 or Shingrix): (1) Any live vaccine, (2) Immunomodulators or immune-suppressive medication, (3) Granulocyte-macrophage colony-stimulating factor, (4) Three or more consecutive days of systemic corticosteroids. Note: subjects on stable-dose steroid replacement (for chronic disease such as iatrogenic deficiency) of prednisone ≤10 mg/day or equivalent are allowed, and (5) Other investigational agents or devices.
* Subjects with active or suspected immunosuppression, immunodeficiency, or autoimmune disease.
* Subjects receiving systemic antiviral therapy.
* Subjects with a positive screening test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or anti-human HIV-1 and 2 antibodies.
* Subjects with a positive screening test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* Subjects with a known history of active or latent tuberculosis (bacillus tuberculosis).

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
SAE Frequency | Day 1 - Day 241
  Frequency of SAEs characterized by type, severity, duration, and relationship to the vaccine (JCXH-105 or Shingrix) recorded from Day 1 post-vaccine administration through follow-up completion
Injection site reaction | 7 days after the first and second vaccination
  Solicited local injection site reactions characterized by frequency, severity, and duration recorded within 7 days after each vaccine administration (JCXH-105 or Shingrix)
Solicited systemic reaction frequency | 7 days after the first and second vaccination
  Solicited systemic adverse reactions characterized by frequency, severity, and duration recorded within 7 days after each vaccine administration (JCXH-105 or Shingrix)
AE frequency | 30 days after the first and second vaccination
  Adverse events (AEs) including unsolicited AEs, characterized by type, severity, duration, and relationship to the vaccine (JCXH-105 or Shingrix) recorded from Day 1 post-vaccine administration to within 30 days following each vaccine administration
Medically attended AE frequency | Day 1 - Day 241
  Medically attended AEs (MAAEs) characterized by frequency, severity, duration, and relationship to the vaccine (JCXH-105 or Shingrix) recorded from Day 1 post-vaccine administration (JCXH-105 or Shingrix) through follow-up completion
The frequency of potential immune-mediated adverse events" | Day 1 - Day 241
  Potential immune-mediated disease (pIMDs) characterized by frequency, severity, duration, and relationship to the vaccine (JCXH-105 or Shingrix) recorded from Day 1 post-vaccine administration (JCXH-105 or Shingrix) through follow-up completion

SECONDARY OUTCOMES:
Cellular immunogenicity of the JCXH-105 and Shingrix vaccine | Day 1 - Day 241
  Frequency of glycoprotein E (gE)-specific CD4+ T cells expressing 2 or more markers of activation in peripheral blood mononuclear cells (PBMCs) analyzed with flow cytometry on Day 1 pre-dose (baseline) and Days 15, 31, 75, 91, and 241 (Follow-up visit)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - CenExel RCA, Hollywood, Florida
  - CenExel FCR, Tampa, Florida
  - CenExel HRI, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: No